CLINICAL TRIAL: NCT02359214
Title: Effect of Vitamin D3 Supplementation on Cardiometabolic Risk Factors in a Cohort of Overweight and Obese Adults in the United Kingdom (UK)
Brief Title: Effect of Vitamin D3 Supplementation on Cardiometabolic Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 855/13/AT/CSN
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Cardiovascular Disease; Diabetes; Bone Disease
Keywords: Vitamin D; Cardiovascular disease; Diabetes; Obesity; Cardiometabolic; Bone disease
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Bone Diseases; Obesity | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 Supplement (Active Comparator): This group will receive a daily dose of 5000IU (125µg) vitamin D3 (which is half of the recommended safe tolerable upper intake level of vitamin D for healthy individuals) for eight weeks.
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): This group will receive 100% lactose placebo daily for eight weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 5000IU (125mcg) vitamin D3 tablet daily over 8 weeks (56 days).
  Other Names: Cholecalciferol
  Arms: Vitamin D3 Supplement
Other: Placebo — 100% Lactose tablet daily over 8 weeks (56 days).
  Other Names: Non-active ingredient
  Arms: Placebo

SUMMARY:
Supplementation studies with vitamin D have been performed where cardiometabolic risk markers have been assessed but these are few, and results are inconsistent. Hence, the purpose of this study is to determine:

1. Whether administering supplemental Vitamin D3 at a dose of 5000IU/day (125µg) in overweight and obese adult participants for 8 weeks will significantly increase circulating concentrations of 25(OH)D or achieve optimal vitamin D status.
2. Whether administering supplemental Vitamin D3 at a dose of 5000IU/day (125µg) in overweight and obese participants for 8 weeks will significantly improve the cardiometabolic parameters measured.
3. To evaluate the relationship between these variables and 25(OH)D concentration. We hypothesise that there will be a significant increase in plasma 25(OH)D following 8 weeks (56days) supplementation of oral vitamin D3 at a dose of 5000IU/day (125µg); Administering supplemental Vitamin D3 at a dose of 5000IU/day (125µg) in overweight and obese participants for 8 weeks will significantly improve the cardio metabolic parameters measured, and there will be a relationship between these variables and 25(OH)D concentrations.

DETAILED DESCRIPTION:
This study is a parallel randomised, double-blind placebo - controlled trial which will be conducted at the University of Chester, Chester, United Kingdom. Ethical permission has been obtained through the University of Chester Faculty Research Ethics Committee(855/13/AT/CSN). Participants, especially students/staff will be recruited from the University of Chester by email, posters/leaflets.

Males were chosen for this study due to their higher risk of developing cardiometabolic diseases compared to premenopausal women. The participants will be randomised to receive either a vitamin D supplement (5000IU (125µg)/d) or placebo for eight weeks. A computer generated random number sequence will be used to assign participants to the intervention and placebo group. Eligibility will be based on 25(OH)D assessment made at a screening visit before the baseline visit, and participants with plasma 25(OH)D level ≤ 75nmol/l will be invited to participate in the study. To ensure compliance with the intervention, participants will be sent reminders about the intervention appointments by email or phone calls. The study will be performed according to the declaration of Helsinki. All participants will provide written consent. Study participants will be instructed to store the study supplements at room temperature. All unconsumed supplements will be returned and counted to assess compliance.

MEASUREMENTS Dietary intake will be estimated at baseline and post intervention using a three day food diary and information about health conditions, medications and health related behaviors will be assessed by a pre-screen test questionnaire, physical activity will be evaluated as the average of the metabolic equivalent of task (MET-min/week) using the International Physical Activity Questionnaire. Participants will be assessed at baseline (day 0), days 28 and 56. The plasma samples will be batch analyzed at the end of the trial.

ANTHROPOMETRIC MEASUREMENTS Height (m2) will be measured without shoes at baseline, using a stadiometer to the nearest 0.1cm precision, Body weight (kg) will be measured without shoes at baseline through post intervention using a digital scale with participants wearing light indoor clothing, BMI will be calculated as weight in kilograms divided by the square of height in meters (kg/m2), and waist circumference at the iliac crest will be measured with a tape measure with the subject standing.

PULSEWAVE VELOCITY AND BLOOD PRESSURE MEASUREMENTS Participants will be given a glass of water and allowed to rest for 5 minutes in a supine position and afterwards the pulse wave velocity meter (Arteriograph) cuff, for measuring arterial stiffness and blood pressure will be placed tightly round the dominant arm. Overall, three measurements will be performed but only the mean of two measurements will be taken.

BIOCHEMICAL MEASUREMENTS A morning blood sample will be collected by venepuncture from the antecubital vein according to standard protocols, with participants in a sitting position after an overnight fast of at least 8 hours. Blood samples will be drawn into 10ml lithium heparin and ethylene diamine triacetic acid (EDTA) tubes to avoid clotting after which they will be immediately transferred into an ice box and then centrifuged for 10 minutes at four degrees Celsius at 3500rpm. Afterwards the centrifuged plasma will be transferred into aliquots and stored at -80 degrees Celsius until analyzed.

CONDUCT OF THE STUDY

This study will require the participants to attend four clinic sessions on four separate days.

Clinic 1(day 0): Participants are expected to complete a consent form and screening test questionnaire after which their weight, height and waist circumference are to be measured. Afterwards, approximately 0.5ml of blood will be collected by finger prick and put in a heparin tube to avoid clotting for vitamin D status screening to ascertain if participant is eligible to partake in the study. Eligible participants will be invited to take part in the study.

Clinic 2 (week 0): Weight, height, waist circumference and blood pressure and body fat measurements will be performed. Afterwards, 25ml of blood will be collected to assess the cardiometabolic risk markers. Participants will then be randomised to receive either vitamin D or placebo (without the active ingredient) supplements for the intervention period.

Clinic 3 (week 4): The procedure performed in clinic 2 will be repeated in this clinic.

Clinic 4 (Week 8): The procedure performed in clinic 2 will be repeated. It is anticipated that the maximum length of each clinic visit will be 45mins.

Participants will be expected to complete a three-day food diary and physical activity questionnaire at Clinic 2 and 4.

SAMPLE-SIZE ESTIMATION

The estimated sample size will be 58 (29 per group), this sample size will allow for the detection of a treatment difference at 95% power, 0.97 effect size and 5% significance. The power calculation was based on a study by (Witham et al., 2012), and the primary outcome flow mediated dilation (FMD) a parameter of endothelial function from which an estimate of 29 per group was obtained, to allow for loss to follow up, sample size was increased to 37 (25%) per group (n= 74). Sample size estimation was conducted using G. Power version 3.1 software.

DATA-ANALYSIS

Data will be checked for a normal distribution by using Shapiro-Wilk since n = 74, and a homogenous variance will be assessed by Levene's statistic. if assumptions of a normal distribution and homogenous variance have been met , a parametric approach will be adopted,if not, a non parametric approach will be adopted

To assess the difference between the groups and the repeated measurement, i will perform a Mixed Model Anova,and any difference observed will be further analysed by a post- hoc, Tukey test.

To check for a relationship between variables and 25(OH)D, Pearson's correlation will be conducted if assumptions were met or spearman's correlation if assumptions were not met .

Descriptive statistics will be consulted to determine where findings differ from baseline values.The mean and standard deviation will provide information about changes that will occur.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18-65 years,
* Those with a BMI ≥ 25kg/m2
* Those with plasma 25(OH)D concentrations < 75nmol/l

Exclusion Criteria:

* Those with gastrointestinal disease, cardiovascular disease, diabetes, osteoporosis, renal and hepatic disorders
* Those taking weight loss drugs
* Those taking cholesterol lowering drugs
* Those currently on a weight reduction programme
* Those with blood pressure ≥ 160/90 mm Hg
* Those taking vitamin D/calcium supplements

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pulsewave Velocity | 0,4 and 8 weeks
  Arterial Stiffness

SECONDARY OUTCOMES:
Aix Brachial | 0,4 and 8 weeks
  Haemodynamic measure
Aix Aortic | 0,4 and 8 weeks
  Haemodynamic measure
Mean Arterial Pressure | 0,4 and 8 weeks
  Haemodynamic measure
Pulse Pressure | 0,4 and 8 weeks
  Haemodynamic measure
Systolic Blood Pressure | 0,4 and 8 weeks
  Haemodynamic measure

OTHER OUTCOMES:
Diastolic Blood Pressure | 0,4 and 8 weeks
  Haemodynamic measure
E-selectin | 0,4 and 8 weeks
  Biomarker
LDL Cholesterol | 0,4 and 8 weeks
  Biomarker
HDL Cholesterol | 0,4 and 8 weeks
  Biomarker
Total Cholesterol | 0,4 and 8 weeks
  Biomarker
Triacylglycerols | 0,4 and 8 weeks
  Biomarker
Plasma Isoprostanes | 0,4 and 8 weeks
  Biomarker
Plasma Renin | 0,4 and 8 weeks
  Biomarker
Plasma C-Reactive Protein (CRP) | 0,4 and 8 weeks
  Biomarker
Plasma Glucose | 0,4 and 8 weeks
  Biomarker
Plasma Insulin | 0,4 and 8 weeks
  Biomarker
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | 0,4 and 8 weeks
  Insulin Resistance
Plasma 25(OH)D | 0,4 and 8 weeks
  Biomarker
Plasma Parathyroid Hormone (PTH) | 0,4 and 8 weeks
  Biomarker
Plasma Osteocalcin | 0,4 and 8 weeks
  Biomarker
Plasma Aldosterone | 0,4 and 8 weeks
  Biomarker
Plasma Angiotensin II | 0,4 and 8 weeks
  Biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Sohail Mushtaq, PhD, Principal Investigator — University of Chester
Locations (1):
- University of Chester, Chester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
I intend to report general participant characteristics, laboratory measurements and details of randomisation in my thesis after writing is complete by February 2017. IPD will possibly be published in nutrition and medical journals by September 2017.

REFERENCES:
- [Derived] Agbalalah T, Mushtaq S. Effect of vitamin D3 supplementation on cardiometabolic disease risk among overweight/obese adult males in the UK: A pilot randomised controlled trial. J Hum Nutr Diet. 2023 Feb;36(1):216-225. doi: 10.1111/jhn.13021. Epub 2022 May 9. PMID 35451536